CLINICAL TRIAL: NCT03560830
Title: START & STOPP in GWI Stress Test Activated Reversible Tachycardia & Stress Test Originated Phantom Perception in Gulf War Illness
Brief Title: START & STOPP in GWI
Acronym: START
Status: Completed | Type: Observational
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, James Baraniuk, MD, Professor of Medicine, Georgetown University
Other Study IDs: 2015-0579
Record Dates: First submitted 2018-04-18; First posted 2018-06-18 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Gulf War Syndrome
MeSH Terms: conditions — Persian Gulf Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum, plasma, and buffy coat were collected before exercise, and 1, 4 and 24 hr after exercise.
  Cerebrospinal fluid was collected after the 2nd exercise stress test Cheek swabs were collected at screening
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control: Sedentary control subjects with no medical or psychiatric disorder
  Interventions: Other: 2 submaximal exercise stress tests
- POTS GWI: GWI with Postural Orthostatic Tachycardia Syndrome (POTS) GWI veterans who had postural orthostatic tachycardia before exercise and after 2 submaximal exercise stress tests. Postural orthostatic tachycardia was defined by 2015 Consensus as an increase in heart rate of greater than or equal to 30 beats per minute between recumbent (after 5 minutes of rest) and standing up. Standing heart rates were measured every minute for 5 minutes. Postural orthostatic tachycardia was defined if the change in heart rate was more than 30 beats per minute at at least 2 of the 5 standing time points. The average change in heart rate did not have to be above 30. There were 11 GWI POTS subjects.
  Interventions: Other: 2 submaximal exercise stress tests
- START: START = Stress Test Activated Reversible Tachycardia One third of GWI veterans were found to have normal changes in heart rate between recumbent and standing (usual change ~10 to 15 beats per minute) BEFORE EXERCISE, but AFTER EXERCISE (submaximal exercise stress tests) they developed postural orthostatic tachycardia with changes in heart rate of 30 or more between recumbent and standing. The effect was transient as it lasted about 36 to 48 hr.
  The START group had brainstem atrophy and reduced brain activation during a cognitive task compared to sedentary control and other GWI subjects.
  Interventions: Other: 2 submaximal exercise stress tests
- STOPP: STOPP = Stress Test Originated Phantom Perception Two thirds of GWI veterans were found to have normal changes in heart rate between recumbent and standing (usual change ~10 to 15 beats per minute) both before and after 2 submaximal exercise stress tests. STOPP did not develop postural orthostatic tachycardia. their changes were equivalent to the sedentary control group.
  The STOPP group increased brain activation of the basal ganglia and anterior insula during a cognitive task compared to sedentary control subjects.
  Interventions: Other: 2 submaximal exercise stress tests

INTERVENTIONS:
Other: 2 submaximal exercise stress tests

SUMMARY:
Gulf War Illness (GWI) veterans were divided into 2 pathophysiological groups based on their orthostatic tachycardia responses after submaximal exercise. Two thirds had normal increases of 10 to 15 beats per minute between recumbent and standing both before and after exercise. These were termed the Stress Test Originated Phantom Perception (STOPP) phenotype. In contrast, one third had increases in heart rate of more than 30 beats per minute indicating that exercise induced postural tachycardia; there were the Stress Test Activated Reversible Tachycardia (START) group. This study aimed to confirm the original findings of Rayhan (2013).

DETAILED DESCRIPTION:
Gulf War Illness (GWI) veterans had heart rate and blood pressure measured lying down, and then for 5 minutes standing up. Before exercise, all GWI had normal changes of 10 to 15 beats per minute upon standing up. Then they had submaximal bicycle exercise stress tests. Rayhan et al. (2013) discovered that two thirds of the subjects had the same, unchanged response of about 10 to 15 beats per minute upon standing both before and after exercise. These were termed the Stress Test Original Phantom Perception (STOPP) phenotype. In contrast, one third of GWI veterans were found to have normal postural changes before exercise, but all the stress tests they had larger changes in heart rate of over 30 beats per minute. They were termed the Stress Test Activated Reversible Tachycardia (START) phenotype.

The importance of the START phenotype was indicated by finding that they had brain stem atrophy by MRI voxel based morphometry, reduced brain blood flow and activation during a cognitive task performed in the fMRI scanner, and differences in biomarkers compared to STOPP and sedentary control subjects.

This study was designed to use the identical exercise protocol to verify or refute the presence of START and STOPP phenotypes in GWI.

The incremental change in heart rate between recumbent and standing (Delta HR) was determined by having subjects lie quietly at rest. Heart rate and blood pressure was measured at 1 minute intervals. The average recumbent heart rate was determined. Then subjects stood up without assistance. Beginning 1 minute after standing up, heart rate was measured at 1 minute intervals for 5 minutes. Delta HR was found by subtracting each of the 5 standing measurements minus the average recumbent heart rate. If a subject had 2 or more Delta HR measurements of 30 beats per minute or greater while standing, they were called Stress Test Activated Reversible Tachycardia (START).

The threshold of 30 beats per minute for Delta HR was based on the criteria for Postural Orthostatic Tachycardia Syndrome (POTS). However, START subjects had normal Delta HR of 10 to 15 before exercise, and so did not have POTS. This was a key finding of the original study that we plan to verify in this study.

Study Design:

Pre-exercise recumbent and standing heart rate measurements and m Magnetic resonance imaging (MRI).

Exercise: Submaximal bicycle exercise stress test. Subjects were monitored while sitting on the bike for 5 minutes. Cycling started with a gradual increase in resistance to increase heart rate to 70% of maximum predicted heart rate (pHR = 220-Age). Cycling continued at 70%pHR for 25 minutes or until the subject wanted to stop. After 25 minutes, the exercise level was increased gradually to reach 85%pHR equivalent to a cardiac stress test. After stopping, heart rate was measured for 5 more minutes while sitting.

Post-Exercise: Recumbent and standing heart rate measurements were performed approximately 3, 8, 24 and 36 hours after exercise. Specific times could not be scheduled because of the timing of MRI scans and other procedures.

Outcome measure: DeltaHR was the difference between standing heart rates minus average recumbent heart rate. Changes in DeltaHR were measured for up to 48 hr after exercise.

START definition: DeltaHR of 30 more greater at 2 or more time points in the 48 hr after submaximal exercise.

ELIGIBILITY:
Inclusion Criteria:

Gulf War Illness subjects: "Kansas" criteria of Lea Steele (2000). Healthy Veterans: Have never met criteria for GWI, Chronic Multisymptom Illness (CMI), or any of the other related conditions.

All subjects: A score of 24 or more on the Mini Mental Status Examination.

Exclusion Criteria:

HIV / AIDS subjects Pregnant women. Active duty military personnel. Children under age of 18 years Incarcerated people (in jail) Cognitive impairment such as mental retardation, severe head injury, stroke, proven multiple sclerosis, "melancholic" suicidal major depression, schizophrenia, dementia, Alzheimer disease, Parkinson's disease, brain injury, severe head injury, bleeding into brain, have been unconscious for more than 1 day (in a coma), seizures, multiple sclerosis, or other serious neurological disease.

Metal implants such as prostheses, wires, plates, or screws that may heat up in the magnetic resonance imaging scanner and cause harm.

Claustrophobia. Abnormal laboratory and questionnaire results. Heart, lung, kidney, arthritis, autoimmune, cancer, and other chronic illnesses, leg amputations, heart attacks (myocardial infarction), coronary artery disease, abnormal heart rhythms, uncontrolled high blood pressure or strokes, lung disease from smoking or other causes, painful, swollen or deformed joints related to arthritis or autoimmune diseases, weakness from nerve damage, liver disease (alcoholic cirrhosis), inflammatory bowel disease (Crohn's disease, ulcerative colitis), or cancer Medications. Drugs that interfere with heart, lung, brain and nerve function Problems Drawing Blood.

Subjects may participate if they have well controlled diabetes or thyroid disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Gulf War Illness subjects had to be in the US military for at least 30 days between August 1, 1990 and July 31, 1991, deployed to the Persian Gulf, and to meet the "Kansas" criteria for Gulf War Illness.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-06-18 (Actual)

PRIMARY OUTCOMES:
START Phenotype | 48 hour
  Delta heart rate (deltaHR) greater than 30 beats per minute within 48 hr of performing submaximal exercise stress test

CONTACTS AND LOCATIONS:
Overall Officials: James N Baraniuk, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
A manuscript is being written to describe the protocol and outcomes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2018-2010
Access Criteria: Open access

REFERENCES:
- [Background] Baraniuk JN, Shivapurkar N. Exercise - induced changes in cerebrospinal fluid miRNAs in Gulf War Illness, Chronic Fatigue Syndrome and sedentary control subjects. Sci Rep. 2017 Nov 10;7(1):15338. doi: 10.1038/s41598-017-15383-9. PMID 29127316
- [Result] Rayhan RU, Washington SD, Garner R, Zajur K, Martinez Addiego F, VanMeter JW, Baraniuk JN. Exercise challenge alters Default Mode Network dynamics in Gulf War Illness. BMC Neurosci. 2019 Feb 21;20(1):7. doi: 10.1186/s12868-019-0488-6. PMID 30791869
- [Result] Garner RS, Rayhan RU, Baraniuk JN. Verification of exercise-induced transient postural tachycardia phenotype in Gulf War Illness. Am J Transl Res. 2018 Oct 15;10(10):3254-3264. eCollection 2018. PMID 30416666
- [Result] Baraniuk JN, Shivapurkar N. Author Correction: Exercise - induced changes in cerebrospinal fluid miRNAs in Gulf War Illness, Chronic Fatigue Syndrome and sedentary control subjects. Sci Rep. 2018 Apr 19;8(1):6455. doi: 10.1038/s41598-018-23238-0. PMID 29674668
- [Result] Rayhan RU, Ravindran MK, Baraniuk JN. Migraine in gulf war illness and chronic fatigue syndrome: prevalence, potential mechanisms, and evaluation. Front Physiol. 2013 Jul 24;4:181. doi: 10.3389/fphys.2013.00181. eCollection 2013. PMID 23898301